CLINICAL TRIAL: NCT04649320
Title: Investigation of the Perception of the COVID-19 Pandemic in Patients With Haematological or Solid Neoplasias Using Patient-reported Outcome Measures (PROMs)
Brief Title: Perception of the COVID-19 Pandemic in Patients With Haematological or Solid Neoplasias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1264/2020
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID19 pandemic; cancer patients; distress; HRQOL
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer patients: adult cancer patients, with solid or hematologic malignancies, neither tested positive nor having COVID19 symptoms
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — 1. 13-item questionnaire about cancer patient's distress and everyday life,
  2. EORTC-QLQ-C30

SUMMARY:
Cancer patients are among the most vulnerable individuals, whose health-related quality of life (HRQOL) may be substantially impacted by the COVID19 pandemic. We want to study how the COVID-19 pandemic influences the life of cancer patients and how these patients cope with the additional distress with the aim to facilitate the development of improved future interventional strategies to maintain resilience and HRQOL

DETAILED DESCRIPTION:
In December 2019, the novel human pathogenic virus "SARS-CoV2" from the coronavirus family was identified, causing a respiratory disease known as "COVID19" (coronavirus disease 2019). COVID19 manifests itself primarily with influenza-like symptoms, but in special cases it can lead to severe conditions such as ARDS (acute respiratory distress syndrome). Compared to other pulmotropic viruses such as the influenza virus, SARS-CoV-2 is associated with a higher contagiousness and mortality.

Haematological and oncological patients are particularly vulnerable due to their advanced age, immunological restrictions in the context of the underlying disease and the treatment modalities (chemotherapy, radiation therapy, ...).

To evaluate the effects of the COVID19 pandemic on the perception of patients with malignant diseases, we aim to record so-called "patient-reported outcomes" (PROs) from patients at the University Hospital of Innsbruck at the Department of Internal Medicine V (Hematology and Oncology) and at the Department for Radiotherapy and Radiation Oncology. We use the validated EORT QLQ-C30 and a specially developed questionnaire for COVID19.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* validated hematological or oncological disease
* informed consent

Exclusion Criteria:

* Age < 18 years
* Insufficient discernment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult cancer patients, with solid or hematologic malignancies, neither tested positive nor having COVID19 symptoms, with an age over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Influence of the COVID-19 pandemic on cancer patient's daily life | single time
  evaluation via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Stauder, M.D., Principal Investigator — Medical University of Innsbruck, Anichstraße 35, A-6020 Innsbruck, Austria
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No